CLINICAL TRIAL: NCT02408796
Title: A 1-Month, Prospective, Multicenter, Open-Label Study of OTO-201 Given as a Single Supra-Tympanostomy Tube Administration for Treatment of Acute Otitis Media With Tympanostomy Tubes in Pediatric Subjects
Brief Title: Open-Label Study of OTO-201 for Treatment of AOMT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otonomy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201-201505
Record Dates: First submitted 2015-03-27; First posted 2015-04-03 (Estimated); Results first posted 2020-09-23 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Acute Otitis Media; AOMT
Keywords: Acute otitis media with tympanostomy tubes
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OTO-201 (Experimental): 6 mg OTO-201
  Interventions: Drug: OTO-201

INTERVENTIONS:
Drug: OTO-201

SUMMARY:
This is a 1-month, prospective, multicenter, open-label study in pediatric subjects with either unilateral or bilateral acute otitis media with tympanostomy tubes (AOMT). Eligible subjects will receive a single dose of 6 mg OTO-201 to the affected ear(s). The study is designed to characterize safety, procedural factors and clinical effect of OTO-201 administered in subjects with AOMT.

ELIGIBILITY:
Inclusion Criteria includes, but is not limited to:

* Subject is a male or female aged 6 months to 17 years, inclusive
* Subject has a clinical diagnosis of acute otitis media with tympanostomy tubes (AOMT)
* Subject's caregiver is willing to comply with the protocol an attend all study visits

Exclusion Criteria includes, but is not limited to:

* Subject has a history of sensorineural hearing loss
* Subject has tympanic membrane perforation other than the surgical tympanostomy tube perforation
* Subject has a history of known immunodeficiency disease

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl LeBel, PhD, Study Chair — Otonomy, Inc.
Locations (5):
- United States (5):
  - Central California Ear, Nose and Throat, Fresno, California
  - South Florida Pediatric Otolaryngology, Fort Lauderdale, Florida
  - Charlotte Eye, Ear, Nose and Throat Associates, Charlotte, North Carolina
  - Charlotte Eye, Ear, Nose and Throat Associates, Matthews, North Carolina
  - Carolina Ear, Nose and Throat, Orangeburg, South Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- OTO-201: 6 mg OTO-201
  OTO-201
Period: Overall Study
Arm/Group | OTO-201
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | OTO-201
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.16 (1.170)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 22
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Ears With Otorrhea (Drainage From the Middle Ear)
Description: Acute otitis media with tympanostomy tubes in place (AOMT) refers to subjects that have ear tubes present, but have a middle ear infection. Otorrhea is fluid drainage from the middle ear. This outcome is assessed during the otoscopic examination of each affected ear (the ear with the infection). All subjects have otorrhea in the affected ear at Baseline and the assessment is done after administering OTO-201 to be sure there is no infection remaining or no new infection.
Time Frame: Day 29
Population: Safety analysis set: All enrolled and treated subjects; subjects could have either unilateral or bilateral (one ear or both ears) acute otitis media with tympanostomy tubes in place (AOMT)
Measure: Count of Units; unit: affected ears
Units Other Than Participants: affected ears
Arm/Group | OTO-201
Number analyzed (Participants) | 39
Number analyzed (affected ears) | 58
affected ears | 8

2. Primary Outcome: Feasibility of Administration Questionnaire
Description: Issues Administering OTO-201 onto the Tympanic Membrane and the Auditory Canal-facing Side of the Tympanostomy Tube (answered "yes")
Time Frame: Day 1
Population: Safety analysis set: All enrolled and treated subjects.
Measure: Count of Units; unit: ears
Units Other Than Participants: ears
Arm/Group | OTO-201
Number analyzed (Participants) | 39
Number analyzed (ears) | 58
ears | 2

3. Secondary Outcome: Number of Ears With no More Otorrhea (Drainage From the Middle Ear)
Description: Acute otitis media with tympanostomy tubes in place (AOMT) refers to subjects that have ear tubes present, but have a middle ear infection. Otorrhea is fluid drainage from the middle ear. This outcome is assessed during the otoscopic examination of each affected ear (the ear with the infection). All subjects have otorrhea in the affected ear at Baseline and the assessment is done 15 days after administering OTO-201 to see if it worked and there is no more drainage from the middle ear.
Time Frame: Day 15
Population: Safety analysis set: All enrolled and treated subjects
Measure: Count of Units; unit: affected ears
Units Other Than Participants: affected ears
Arm/Group | OTO-201
Number analyzed (Participants) | 39
Number analyzed (affected ears) | 58
affected ears | 50

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | OTO-201
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 23/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OTO-201 (N=39)
Pyrexia (General disorders) | 9
Device Extrusion (General disorders) | 4
Sinusitis (Infections and infestations) | 3
Otitis Media (Infections and infestations) | 2
Otitis Media Acute (Infections and infestations) | 2
Pharyngitis Streptococcal (Infections and infestations) | 2
Diarrhea (Gastrointestinal disorders) | 2
Seasonal Allergy (Immune system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication subject to Sponsor consent.